CLINICAL TRIAL: NCT03778801
Title: Evaluation of Kinesiophobia and Physical Activity Levels in Patients With Fibromyalgia Syndrome and Chronic Neck Pain
Brief Title: Kinesiophobia in Patients With Fibromyalgia Syndrome and Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dr. Melek Aykut Selçuk, Principal Investigator, Aksaray University Training and Research Hospital
Other Study IDs: 2018/155
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia; Neck Pain; Healthy
Keywords: kinesiophobia; physical activity; disability
MeSH Terms: conditions — Fibromyalgia; Neck Pain; Kinesiophobia; Motor Activity | interventions — Pain Measurement; Disability Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- fibromyalgia syndrome: Thirty patients with a diagnosis of fibromyalgia syndrome according to the 2016 revised American College of Rheumatology Fibromyalgia Syndrome diagnostic criteria and a disease duration of longer than three months
  Interventions: Diagnostic Test: kinesiophobia
- chronic neck pain: 30 patients with chronic neck pain lasting for more than three months and didn't meet 2016 revised American College of Rheumatology Fibromyalgia Syndrome diagnostic criteria.
  Interventions: Diagnostic Test: kinesiophobia
- healthy controls: 30 healthy controls without pain or additional disease
  Interventions: Diagnostic Test: kinesiophobia

INTERVENTIONS:
Diagnostic Test: kinesiophobia — The investigators assessed pain intensity, kinesiophobia, fatigue, depression, physical activity level and disability in patients with fibromyalgia syndrome and chronic neck pain, and healthy individuals in this cross-sectional study.
  Other Names: physical activity level; pain intensity; disability; fatigue; depression

SUMMARY:
Kinesiophobia which is described as fear of movement reduces physical activity levels and increases the risk of chronic pain. The investigators consider that kinesiophobia levels are higher in patients with fibromyalgia syndrome and chronic neck pain so that physical activity levels are lower in this patient groups. Because there are not enough studies, the investigators aimed to evaluate kinesiophobia and physical activity levels in this patients.

DETAILED DESCRIPTION:
Objective: To evaluate pain, kinesiophobia, physical activity, depression, disease severity, and fatigue in patients with fibromyalgia syndrome or chronic neck pain and healthy controls.

Design: Cross-sectional study. Setting: Tertiary Health Care Center, Aksaray, Turkey Participants: 30 patients with fibromyalgia syndrome (Group 1), 30 patients with chronic neck pain (Group 2), and 30 healthy individuals (Group 3) were included.

Main Outcome Measures: Outcome measures were Visual Analogue Scale (VAS)-pain and fatigue, Tampa Scale of Kinesiophobia (TSK), Beck Depression Inventory (BDI), International Physical Activity Questionnaire (IPAQ) Short Form, Fibromyalgia Impact Questionnaire (FIQ), Neck Pain Disability Index (NPDI).

ELIGIBILITY:
Inclusion Criteria:

Participants with a clinical diagnosis of fibromyalgia syndrome Participants with a clinical diagnosis of chronic neck pain Healthy participants Participants with fibromyalgia syndrome and chronic neck pain has had a disease duration more than three months

Exclusion Criteria:

Malignant disease Systemic infectious disease Rheumatic disease Operation Pregnancy Psychological or cognitive disorder History of physical therapy within the last three months History of intra-articular or intra-ligamentary injection within the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients were recruited from a physical medicine and rehabilitation outpatient clinic of Aksaray University Training and Research Hospital, Aksaray, Turkey. The healthy control group was consisting of doctors, nurses, medical secretaries who work in Aksaray University Training and Research Hospital, and patient care providers that have no pain and additional diseases
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melek A Selçuk, Principal Investigator — Aksaray University Training and Research Hospital
Locations (1):
- Aksaray University Training and Research Hospital, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from a physical medicine and rehabilitation outpatient clinic of Aksaray University Training and Research Hospital, Aksaray, Turkey. The healthy control group was consisting of doctors, nurses, medical secretaries who work in Aksaray University Training and Research Hospital, and patient care providers that have no pain
Period: Overall Study
Arm/Group | Fibromyalgia Syndrome | Chronic Neck Pain | Healthy Controls
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibromyalgia Syndrome | Chronic Neck Pain | Healthy Controls | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 90
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.96 (10.88) | 38.50 (11.65) | 35.40 (9.95) | 38.91 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 22 | 77
  Male | 2 | 3 | 8 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Tampa Scale of Kinesiophobia
Description: Based on a four-point Likert type, this scale contains 17 items that evaluate fear and anxiety related to physical activity. A total score of greater than 37 is accepted as statistically significant and interpreted as a high level of kinesiophobia. Minimal and maximal scores could be between 17-68 points. Higher scores indicate higher levels of kinesiophobia.
Time Frame: 4-8 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia Syndrome | Chronic Neck Pain | Healthy Controls
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 41.70 (6.30) | 38.33 (7.98) | 30.83 (8.84)

2. Primary Outcome: International Physical Activity Questionnaire Short Form
Description: This questionnaire consists of seven items that measure the duration of the participants' physical activity, walking and sitting within the last seven days in the metabolic equivalent (MET)-min/week unit. 3 or more days of vigorous activity of at least 20 minutes per day or 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day or 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-minutes/week are proposed to be moderate level. Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/week or 7 or more days of any combination of walking, moderate- or vigorous-intensity activities accumulating at least 3000 MET-minutes/week are proposed to be high level. Some activity is reported but not enough to meet categories of moderate or high levels, it is proposed to be low level.
Time Frame: 5-10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Fibromyalgia Syndrome | Chronic Neck Pain | Healthy Controls
Number analyzed (Participants) | 30 | 30 | 30
Participants
  low | 21 | 14 | 7
  moderate | 7 | 11 | 16
  high | 2 | 5 | 7

3. Primary Outcome: Beck Depression Inventory
Description: This is a 21-item questionnaire that investigates the characteristic attitudes and symptoms of depression. A score of 10 or higher indicates depression. Minimal and maximal scores can be 0-63 points. Higher scores indicate higher levels of depression.
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia Syndrome | Chronic Neck Pain | Healthy Controls
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 18.37 (8.07) | 12.03 (7.09) | 5.44 (5.68)

4. Primary Outcome: Fibromyalgia Impact Questionnaire
Description: Fibromyalgia Impact Questionnaire aims to evaluate the arthritis symptoms and functional status of patients with fibromyalgia syndrome through 21 questions that inquire about physical functions, work-related situations, depression, anxiety, waking up tired, pain, stiffness, and fatigue. Higher scores indicate greater impact of fibromyalgia on functioning. Final score should range from 0 to 80.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia Syndrome | Chronic Neck Pain | Healthy Controls
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 49.79 (22.60) | 44.44 (15.71) | 13.79 (10.17)

5. Primary Outcome: Neck Pain Disability Index
Description: This index consists of 20 questions that assess severity of neck pain and the extent to which the pain affects the social, professional and daily activities of patients.Final score should range from 0 to 100. Higher scores indicate greater levels of disability.
Time Frame: 5-8 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Chronic Neck Pain: 30 patients with chronic neck pain lasting for more than three months
Arm/Group | Chronic Neck Pain | Healthy Controls
Number analyzed (Participants) | 30 | 30
score on a scale | 49.06 (21.65) | 6.16 (10.21)

6. Primary Outcome: Visual Analog Scale for the Evaluation of Pain
Description: For this evaluation, the patient is asked to mark his/her severity of pain on a horizontal 100-mm line with 0 on one end representing no pain and 100 on the other end represent very severe pain. Higher scores indicate higher levels of pain intensity.
Time Frame: 0.5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia Syndrome | Chronic Neck Pain | Healthy Controls
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 75.83 (27.26) | 50.33 (23.85) | 0 (0)

7. Primary Outcome: Visual Analog Scale for the Evaluation of Fatigue
Description: For this evaluation, the patient is asked to mark his/her severity of fatigue on a horizontal 100-mm line with 0 on one end representing no fatigue and 100 on the other end represent very severe fatigue.
Time Frame: 0.5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fibromyalgia Syndrome | Chronic Neck Pain | Healthy Controls
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 74.66 (28.37) | 64.33 (24.59) | 41.66 (23.05)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed
Description: Adverse Events were not monitored/assessed
Arm/Group | Fibromyalgia Syndrome | Chronic Neck Pain | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small sample size, presence of a difference between the fibromyalgia syndrome and control groups in terms of age and gender, and lack of Neck Pain Disability Index evaluation in the fibromyalgia syndrome group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03778801/Prot_SAP_001.pdf